CLINICAL TRIAL: NCT01969578
Title: A Randomized Phase II Study to Evaluate the Efficacy and Safety of Chemotherapy (CT) vs Androgen Deprivation Therapy (ADT) in Patients With Recurrent and/or Metastatic, Androgen Receptor (AR) Expressing, Salivary Gland Cancer (SGCs)
Brief Title: Androgen Deprivation Therapy in Advanced Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1206; 2013-000314-38 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-10-25 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Salivary Gland Cancer
Keywords: salivary duct cancer; adenocarcinoma, NOS; androgen deprivation; androgen receptor
MeSH Terms: conditions — Salivary Gland Neoplasms; Adenocarcinoma; Bulbo-Spinal Atrophy, X-Linked | interventions — bicalutamide; Triptorelin Pamoate; Cisplatin; Doxorubicin; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Active Comparator): Chemotherapy = either Cisplatin + Doxorubicin or Carboplatin + Paclitaxel
  Patients from cohort A (chemonaïve) may be randomized in this arm to receive chemotherapy
  Interventions: Drug: Cisplatin + Doxorubicin; Drug: Carboplatin + Paclitaxel
- Androgen Deprivation Therapy (ADT) (Experimental): ADT = bicalutamide + triptorelin
  Patients from cohort A (chemonaive) may be randomized to receive ADT, and patients from cohort B (pre-treated) will receive ADT without having been randomized.
  Interventions: Drug: bicalutamide + triptorelin

INTERVENTIONS:
Drug: bicalutamide + triptorelin
  Arms: Androgen Deprivation Therapy (ADT)
Drug: Cisplatin + Doxorubicin
  Arms: Chemotherapy
Drug: Carboplatin + Paclitaxel
  Arms: Chemotherapy

SUMMARY:
Salivary Gland (SG) Cancers are a rare and heterogeneous group of tumors, usually approached by multidisciplinary teams in high specialized centers. Until today no standard of care exists to treat these cancers. The identification of a target, the androgen receptor, in SG tumors has allowed for new treatment strategies options for this rare group of diseases. As a matter of fact, strong positivity for androgen expression has been found in salivary duct carcinoma and adenocarcinomas. The purpose of this study is therefore to evaluate the efficacy and safety of chemotherapy versus androgen deprivation therapy (ADT) in patients with recurrent and/or metastatic AR expressing SGCs.

The study will include two cohorts of patients: Cohort A, which comprises chemo-naïve patients, and Cohort B, which comprises pretreated patients.

DETAILED DESCRIPTION:
Patients in Cohort A will be randomized 1:1 at the study entry to receive ADT (triptorelin + bicalutamide 50 mg) or standard chemotherapy. Patients of Cohort A randomized to the control arm (chemotherapy arm) will be given the option to enter Cohort B at the time of disease progression. As long as Cohort A is open to recruitment, patients who will be treated by chemotherapy will be simultaneously enrolled in Cohort B. Accrual in Cohort B will be stopped when recruitment of 76 eligible patients in Cohort A is reached.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of recurrent and/or metastatic salivary duct cancer; adenocarcinoma, NOS; and AR expression in at least 70% of nuclei of neoplastic cells based on central review
* Sufficient tissue must be available either historically or a biopsy must be done as a part of this study and sent to central review for patients enrolled in both cohorts
* Presence of at least one uni-dimensional measurable lesion by CT-scan or MRI according to RECIST criteria version 1.1 (target lesion).
* Patients older than 18 years old;
* Performance Status ECOG 0-1;
* Adequate bone marrow function:
* WBC ≥ 3.5/10exp9L
* absolute neutrophil count ≥ 1,5x10exp9/L
* hemoglobin > 9 g/dL
* platelet count ≥ 100x10exp9/L
* Adequate liver function:
* AST < 2.5 times upper limit of normal
* ALT < 2.5 times upper limit of normal
* bilirubin < 1.5 times upper limit of normal
* the concomitant evidence of AST < 2.5 times upper limit of normal, ALT < 2.5 times upper limit of normal and bilirubin > 1.5 times upper limit of normal is not allowed
* Adequate renal function:
* serum creatinine level (≤ 1.3 mg/dL)
* calculated creatinine clearance ≥ 60 mL/min based on the standard Cockcroft and Gault formula
* Adequate cardiac function as demonstrated by a clinically normal 12 lead ECG; additionally for patients who will receive Cisplatin and Doxorubicin adequate cardiac function should be demonstrated by a left ventricular ejection fraction (LVEF) ≥ 50% (within 2 weeks prior to treatment start)

Exclusion Criteria:

* Actively bleeding tumor if the patient is intended to be treated with carboplatin
* Patients with bone disease or brain disease as the sole disease site; brain metastases are allowed in case of systemic disease, but must have been treated at least 4 weeks before enrollment and must be stable after that;
* recent history of congestive heart failure, unstable angina within the past 3 months, cardiac arrhythmia, myocardial infarction, congenital long QTc prolongation, stroke, TIA within the past 6 months;
* previous cardiac toxicity induced by another anthracycline or previous exposure to maximum cumulative dose of another anthracycline if the patient is intended to be treated with doxorubicin
* history of allergic reactions attributed to compounds of similar chemical or biological composition to cis/carboplatin, paclitaxel, doxorubicin, bicalutamide or triptorelin;
* concomitant medications with terfenadine, astemizole, cisaprid
* use of phenytoin
* Patients who received vaccine for yellow fever
* active second malignancy during the last five years except non melanomatous skin cancer or carcinoma in situ of the cervix;
* positive serum pregnancy test within 1 week prior to the first dose of study treatment for Women of child bearing potential (WOCBP);
* no adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment for patients of childbearing / reproductive potential.
* psychological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* written informed consent not given according to ICH/GCP, and national/local regulations, before patient registration
* participation in another interventional clinical trial in the preceding 4 weeks prior to randomization
* for cohort A patients: previous chemotherapy for recurrent/metastatic disease (previous chemotherapy given concomitantly with RT in the past is allowed, including cisplatin but it should be completed at least 6 months before enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 37 months after First Patient In
  PFS is a primary outcome for cohort A
Response rate (RR) | 37 months after First Patient In
  RR is a primary outcome for cohort B

SECONDARY OUTCOMES:
Response Rate (RR) | 37 months after First Patient In
  RR is a secondary outcome for cohort A
Progression Free Survival (PFS) | 37 months after First Patient In
  PFS is a secondary outcome for cohort B

OTHER OUTCOMES:
Overall Survival (OS) | 37 months after First Patient In
Adverse Events according to CTCAE v4.0 | 37 months after First Patient In
  adverse events will be recorded using International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI; Kevin Harrington, Study Chair — The Royal Marsden
Locations (26):
- Medical University Vienna - General Hospital AKH, Vienna, Austria
- Belgium (5):
  - ZNA Middelheim, Antwerp
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (9):
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Nantes
  - CHU de Nantes - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Assistance Publique - Hopitaux de Paris - Hopital Tenon, Paris
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Jena-Radiation Therapy and Radiooncology Clinic, Jena
  - Universitaetsklinikum Leipzig-Ambulanzen/Sprechstunden, Leipzig
- Athens University - Attikon University General Hospital, Athens, Greece
- National Institute Of Oncology, Budapest, Hungary
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Provinciale per i Servizi Sanitari - Ospedale Santa Chiara, Trento
- Netherlands (3):
  - Spaarne Gasthuis - Vrije Universiteit Medisch Centrum, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud University Medical Center Nijmegen, Nijmegen